CLINICAL TRIAL: NCT06126302
Title: Analyzing the Changes in Eye Axis Length and Corneal Curvature in Central China From the Perspective of Birth Year
Brief Title: Analyzing the Changes in Eye Axis Length and Corneal Curvature in Central China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Min Ke (Other)
Responsible Party: Sponsor-Investigator, Min Ke, Department of ophthalmology, Zhongnan Hospital, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Other Study IDs: 20231105
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Birth Year-dependent Eye Parameters Change
Keywords: Eye axial length; Corneal curvature; Birth year-dependent

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Before 1930: the patients were divided into ten groups according to the decade of their birth: before 1930
  Interventions: Other: Birth year
- 1930-1939: the patients were divided into ten groups according to the decade of their birth: 1930-1939
  Interventions: Other: Birth year
- 1940-1949: the patients were divided into ten groups according to the decade of their birth: 1940-1949
  Interventions: Other: Birth year
- 1950-1959: the patients were divided into ten groups according to the decade of their birth: 1950-1959
  Interventions: Other: Birth year
- 1960-1969: the patients were divided into ten groups according to the decade of their birth: 1960-1969
  Interventions: Other: Birth year
- 1970-1979: the patients were divided into ten groups according to the decade of their birth: 1970-1979
  Interventions: Other: Birth year
- 1980-1989: the patients were divided into ten groups according to the decade of their birth: 1980-1989
  Interventions: Other: Birth year
- 1990-1999: the patients were divided into ten groups according to the decade of their birth: 1990-1999
  Interventions: Other: Birth year
- 2000-2009: the patients were divided into ten groups according to the decade of their birth: 2000-2009
  Interventions: Other: Birth year
- after 2009: the patients were divided into ten groups according to the decade of their birth: after 2009
  Interventions: Other: Birth year

INTERVENTIONS:
Other: Birth year — we divided the patients according to patients' birth year

SUMMARY:
The Chinese lifestyle has undergone dramatic changes over the past century. In recent years, limited studies reported the changing trend in crucial eye parameters of people born in different decades. This multicenter study analyzed the axial length and average corneal curvature data from patients of four hospital. The trends in the axial length and corneal curvature will be observed.

DETAILED DESCRIPTION:
The Chinese lifestyle has undergone dramatic changes over the past century. In recent years, limited studies reported the changing trend in crucial eye parameters of people born in different decades. This multicenter study analyzed the axial length and average corneal curvature data between 2012 and 2023. There were four clinical centers involved in this study. The study was approved by the Medical Ethics Committee of Zhongnan Hospital, Wuhan University, Yichang center hospital, Jingzhou center hospital , Yichang center hospital and Xiaogan center hospital, and conformed to the tenets of the Declaration of Helsinki. We divided the participants into ten groups of 10 years each based on their year of birth (called birth decade) and observed the trends in the axial length and corneal curvature in different groups.

ELIGIBILITY:
Inclusion Criteria:

- Eligible patients were those aged ≥7 years and who underwent intraocular lens (IOL) Master (version 5.5) biometry for routine examination of cataract or refractive examination (ametropia and presbyopia) between April 2012 and November October 2023. Only patients who would cooperate with examinations to ensure stable and repeatable data (AL was measured 5 times or more, CC was measured 3 times or more, and the coefficient of variation of the measured results were≤15%a coefficient of variation ≤15% was considered low variation) were selected.

Exclusion Criteria:

- Severe systemic disease, corneal diseases, severe dry eyes, serious fundus disease, noticeable lesions of the refractive stroma, inability to cooperate, or poor measurement quality (coefficient of variation> 15%) were the exclusion criteria.

Ages: 7 Years to 130 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients were those aged ≥7 years and who underwent intraocular lens (IOL) Master (version 5.5) biometry for routine examination of cataract or refractive examination (ametropia and presbyopia) between April 2012 and November October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Eye Axial Length | 2023/10
  The Axial length of all patients were measured using the IOL Master 5.5 (Carl Zeiss Meditec, Dublin, CA) biometry system for routine examination of cataracts or refractive examination (ametropia and presbyopia).AL was measured as the distance from the tear film to the retinal pigment epithelium. The mean of 5 measurements wasas taken for final analyses.
Corneal Curvature | 2023/10
  The corneal curvature of all patients were measured using the IOL Master 5.5 (Carl Zeiss Meditec, Dublin, CA) biometry system for routine examination of cataracts or refractive examination (ametropia and presbyopia). Corneal curvature was measured in two meridians: flat keratometry (K1) and steep K (K2). The K value was the mean of K1 and K2. Corneal curvature was measured at least three times. In case of variations in values, measurements were repeated until reproducible results were obtained.

IPD SHARING:
Plan to Share IPD: No